CLINICAL TRIAL: NCT00789945
Title: The Importance of Insulin Timing in Type 1 Diabetes
Brief Title: Timing of Insulin Before Meals Everyday
Acronym: TIME
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: This research was completed before January 18, 2017, and does not meet the ACT requirement to register and report results per the guidance provided in "Clinical Trials Registration and Results Information Submission" dated 09/21/2016.
Sponsor: University of New Mexico (Other)
Collaborators: American Diabetes Association (Other)
Responsible Party: Principal Investigator, David S. Schade, MD, University of New Mexico
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: 08-147
Record Dates: First submitted 2008-11-11; First posted 2008-11-13 (Estimated); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Type 1 Diabetes
Keywords: type 1 diabetes; continuous glucose monitoring; Intensive Insulin therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Study Arm A (Placebo Comparator): Study Arm A will be the primary control arm.
  Interventions: Other: Control
- Study Arm B (Experimental): Study Arm B will serve as the intervention arm.
  Interventions: Other: Study Arm B

INTERVENTIONS:
Other: Control — Study Arm A will consist of patients with Type 1 diabetes who will continue their current intensive insulin therapy regimen with no additional interventions by the investigators. Their primary care providers will continue to manage their diabetes to obtain the best control as possible of their glucose, lipids, and blood pressure. Continuous Glucose Monitoring will be monitored. No timing of premeal insulin administration will be utilized in this arm.
  Other Names: Control group- No "timing" insulin administartion.
  Arms: Study Arm A
Other: Study Arm B — Study Arm B will include participants with type 1 diabetes which will utilize "Timing" to adjust their pre-meal insulin dosages. Participants will continue taking their current insulin and will be placed on a continuous glucose monitor.
  Other Names: Intervention- "Timing" of insulin administration.
  Arms: Study Arm B

SUMMARY:
The inclusion of "Timing of premeal insulin administration (Timing)" in an Intensive Insulin Therapy regimen will reduce A1C by an average of 1% in type 1 diabetic patients who have initial A1C's between 7.0% and 9.0%.

DETAILED DESCRIPTION:
Data:

The Rationale for Timing of the premeal insulin administration - In type 1 diabetes, very little, if any, endogenous insulin is available to handle the carbohydrate load which very rapidly enters the circulation after the start of a meal. In non-diabetic individuals, a complex array of physiological events occurs prior to eating (often called the cephalic phase of insulin secretion) which prepares the pancreas for immediate release of preformed insulin when any meal related increase in blood glucose occurs. This rapid insulin secretion prepares the tissues (primarily muscle and liver) to take up glucose very rapidly and thereby prevent severe hyperglycemia in the postprandial state. Since significant absorption of all short acting insulins (e.g. insulin Lispro, Aspart, or Glulisine) from the subcutaneous tissue does not occur for 15 minutes following injection (26), this delay often results in postprandial hyperglycemia. If the patient happens to be hypoglycemic prior to the meal, this delay can be advantageous, but if he/she is hyperglycemic, then severe postprandial hyperglycemia may result. A rationale solution to this problem would be to time the short acting insulin injection based on the premeal blood glucose, but aside from our one pilot study addressing this strategy, no clinical study has been published supporting this approach. Our grant application is designed to correct this deficiency and provide the scientific data to support this addition to intensive insulin therapy.

We studied the effect of Timing a fixed dose of rapid acting insulin Lispro (Humalog™) in twelve type 1 diabetic subjects who were all made hyperglycemic prior to a standardized diabetic meal (11). In all studies, the dose of insulin of 0.15U/kg (~10 units) remained constant and represented a typical dose utilized by type 1 diabetic patients prior to an evening meal. Each of the twelve diabetic volunteers participated in all four study arms (48 total studies). The insulin Lispro was given at the following times: 1) 30 minutes prior to meal time (-30 minutes), 2) 15 minutes prior to the meal time (-15 minutes), 3) at the meal (0 minutes), and 4) 15 minutes after the meal was begun (+15 minutes). As is shown in Figure 1, a normal postprandial glucose excursion was observed when the insulin was taken 15 minutes prior to the meal. No postprandial excursion was observed when the insulin was taken 30 minutes prior to the meal. This is the desirable outcome in a hyperglycemic individual. Of particular interest is the fact that when the insulin :Lispro was taken right at mealtime (which is the most common pattern in type 1 diabetic patients), significant postprandial hyperglycemia was observed. Figure 2 provides the integrated postprandial glucose excursion (above and below baseline) over the entire 5½ hour study and reflects the data in Figure 1. This study strongly supports the injection of insulin Lispro at least 15 minutes prior to the meal when premeal hyperglycemia is present.

To be certain that the absorption of insulin Lispro was not different between the four studies which might account for the difference in postprandial glucose excursion; we measured free insulin levels during all four research studies. As is shown in Figure 3, when the insulin excursion concentrations are superimposed on each other for each study, no difference in insulin absorption occurred between the four insulin administration protocols. This data strongly supports the concept that timing of the insulin injection prior to the meal has a major effect on glucose kinetics following a meal. Utilization of Timing in an Intensive Insulin Therapy regimen should have a major beneficial effect of suppressing postprandial hyperglycemia and reducing A1C.

Study Design:

The proposed study will be a double-blind, randomized controlled trial of approximately eight months duration per patient. The volunteers will be screened and then randomized to either a Timing protocol (continuing with their Intensive Insulin Therapy regimen) or continuing their usual Intensive Insulin Therapy. All volunteers will utilize Continuous Glucose Monitoring every other month in order to provide data on the magnitude of postprandial hyperglycemia and the incidence of hypoglycemia.

Insulin Timing Algorithm:

Based on our preliminary data (24), we will utilize the following algorithm to time the premeal insulin administration dose: 1) premeal blood glucose >250 mg/dl = take insulin 30 min before the meal, 2) premeal blood glucose between 250 and 150 mg/dl = take insulin 15 minutes before the start of the meal, 3) premeal blood glucose between 150 and 75 mg/dl = take insulin at the start of the meal, and 4) premeal blood glucose < 75 = take insulin 15 min after the start of the meal. Participants will remain on their current insulin to determine if the timing algorithm is indeed effective. The advantages of this algorithm are that it is very easy to remember and practical for the typical patient with type 1 diabetes. It is designed to keep the glucose between 100 mg/dl and 150 mg/dl. It will reduce the postprandial glucose excursion when most needed, i.e. when the premeal glucose is abnormally high and prevent hypoglycemia when the premeal glucose is low.

Statistical Assessment

Power Analysis:

Our pilot data are the only data available in the literature that assesses the effect of timing of the pre-prandial short acting insulin dose. As detailed above, this pilot study was short term so did not include any assessment of changes in A1C. Since A1C is the primary endpoint in the proposed study, we had to estimate the change in A1C that would have occurred with the changes we observed in the integrated postprandial excursion (figure 1 above). Assuming that the postprandial glucose excursion is responsible for 50% of the A1C value (above the normal concentration of 5.5%) as has been estimated in type 1 diabetic patients (16,17), then the variance and mean change in integrated glucose excursion was used to estimate the change in A1C that would be expected in the proposed study. From this data, we calculated that an improvement of A1C of 1% (the difference in A1C between the control Arm A and the intervention Arm B would require 16 subjects per group to provide a power of 90% to detect this difference at a p<0.01. In order to control for a maximum dropout rate of 20%, we will recruit and randomize a total of 40 volunteers for each group (a total of 80 subjects).

Data Analysis:

The primary endpoint for this study will be the difference in A1C levels between experimental Arm A (volunteers not utilizing Timing ) and Group B (volunteers utilizing Timing). This comparison will provide the net effect of Timing and the direct measure of the change in postprandial hyperglycemia. In addition, several sub analyses will be done. This comparison will control for any positive effects that Continuous Glucose Monitoring may have on A1C. In addition, we will integrate the area under the five-hour postprandial glucose curve as provided each day by the Continuous Glucose Monitoring Data for the primary meal of the day (as stated by the patient - usually supper). This data will provide a mechanism of any improvement in A1C observed. Finally, as an indirect assessment of changes in postprandial hyperglycemia, changes in 1, 5-anhydroglucitol (Glycomark™) will be measured every month. We will utilize an "intention to treat analysis" to analyze the data obtained. Analysis of data will be done using NCSS computer software (42).

Clinical Importance:

If our pilot study is validated by the proposed randomized clinical trial in this grant application, a new parameter for control of postprandial glucose will become available for the patient with type 1 diabetes. To date, this concept has not been utilized by healthcare providers because no one has demonstrated that Timing will result in a reduction of A1C. Our proposed grant application is designed to obtain the data that will make the use of Timing an integral part of a glucose control algorithm. Our results are not restricted to type 1 diabetic patients who utilize insulin Lispro since all of the short acting insulin analogs exhibit approximately the same absorption insulin profile (26), Participants will remain on their current insulin regimen. If our hypothesis is proved correct, i.e., that the correct Timing of the premeal insulin bolus will reduce the A1C by an average of 1% in type 1 diabetic individuals with A1Cs between 7.0% and 9.0%, then according to data generated by the Diabetes Control and Complications Trial, a significant reduction in the microvascular and macrovascular complications of diabetes will occur. In addition, the successful completion of this study will provide a stimulus to examine the Timing of premeal insulin in other groups of diabetic patients, including type 2 diabetic patients on insulin therapy, pregnant women with gestational diabetes, and children with type 1 diabetes. Finally, in this day and age of continuing increases in health care costs, the inclusion of Timing will not add any additional financial cost to the diabetic patient's intensive insulin therapy regimen.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetic participants, History of insulin dependance for at least one year, A1C 7%-9%, normal CBC, Chemistry Profile,be sufficiently stable.

Exclusion Criteria:

* pregnant women, children, prisoners, mentally ill individuals, patients currently utilizing continuous glucose monitors.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2008-12 (Actual); Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
To determine the changes in A1C. | 8 months

SECONDARY OUTCOMES:
To determine changes in postprandial glucose excursion during the meal's 5 hour postprandial period. | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: David S Schade, MD, Principal Investigator — University of New Mexico, Health Sciences Center
Locations (2):
- United States (2):
  - UNM HSC Diabetes Research and Treatment Center, Albuquerque, New Mexico
  - Unm Hsc Gcrc, Albuquerque, New Mexico